CLINICAL TRIAL: NCT05529095
Title: Open Label and Placebo-Controlled Assessment of Sublingual Apomorphine (Kynmobi) as Adjunct Therapy for Patients With Refractory Restless Legs Syndrome
Brief Title: Sublingual Apomorphine in Refractory Restless Legs Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: William Ondo, MD (Other)
Collaborators: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor-Investigator, William Ondo, MD, Principal Investigator, The Methodist Hospital Research Institute
Organization: The Methodist Hospital Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO00033518
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Restless Legs Syndrome
Keywords: Refractory
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sublingual Apomorphine (Kynmobi) (Experimental): Sublingual apomorphine to be titrated after initial dose of 10 mg. Titration is dependent on subjects response.
  Interventions: Drug: Apomorphine Sublingual Film
- Placebo (Placebo Comparator): At week 4, subjects will be given randomization packet including 2 drug doses and 2 placebos.
  Interventions: Drug: Apomorphine Sublingual Film; Drug: Placebo

INTERVENTIONS:
Drug: Apomorphine Sublingual Film — Sublingual Apomorphine initial dose 10 mg, titrated depending on symptomatic response.
  Other Names: Kynmobi
Drug: Placebo — Placebo (sugar pill)
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
This is an open label, short placebo-controlled trial in Restless Legs Syndrome (RLS) patients inadequately treated with standard therapy. Investigators hypothesize that the study drug, sublingual apomorphine (Kynmobi), may improve RLS breakthrough symptoms. This study is designed to determine if sublingual apomorphine improves breakthrough symptoms in RLS patients, in addition to subjective responses.

DETAILED DESCRIPTION:
This is an open label, with a short placebo-controlled portion trial using sublingual apomorphine (Kynmobi) in RLS patients inadequately treated with standard therapy, defined by an IRLS > 15 and report of breakthrough symptoms.

At the initial visit, subjects will undergo all baseline and exploratory assessments and be given their first drug dose of 10 mg. They will be monitored for 60 minutes after dose. Subjects orthostatic blood pressure will be taken before ingestion, then 10, 20, 30, and 45 minutes after ingestion. Over the next 4 weeks, subjects will titrate Kynmobi to find optimal dose. Subjects will be instructed to take at least 2 doses before determining if further titration is needed.

At week 4, subjects will return for exploratory assessments. Subjects will be given a randomized study drug packet containing 2 placebos and 2 drug doses. Subjects will be told that 0-4 doses may be placebo or drug. Subjects will have 4 weeks to complete randomization doses. It is anticipated subjects will complete randomization sooner, so they will be given 23 doses of study drug (1 dose per 24 hours for 23 extra days until next visit).

At week 8, subjects will return for exploratory assessments and be given an additional 74 dosed strips. They will return at week 16 for a final visit and undergo exploratory assessments, followed by a safety call two weeks later.

From weeks 0-8, subjects are able to continue their scheduled RLS medications. From weeks 8-16, subjects may make changes to their RLS medications as mutually agreed upon with investigator.

Several questionnaire assessments will be conducted throughout the study to monitor subjects. Subjects will complete the International RLS Rating Scale (IRLS), Restless Legs Syndrome - 6 Scale (RLS - 6), RLS Quality of Life Questionnaire (RLSQoL), RLS Augmentation Scale, Fatigue Severity Scale (FSS), Hamilton Depression Scale (HDS), Clinical Global Impressions (CGI), and Clinical Global Impressions-Change (CGI-C).

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic RLS diagnosed by standard criteria, with an IRLS > 15 while taking at least 1 RLS medication
* Stable RLS medications for at least 2 weeks prior to study entry

Exclusion Criteria:

* Concurrent untreated sleep disorders, not felt to be able stable
* Subjects with any significant, unstable cardiovascular, liver, lung, renal. psychiatric, or neurological diseases (not including RLS)
* Any medical or psychiatric comorbidity that, in the opinion of the investigator, would make study compliance difficult to achieve
* Intravenous iron within 4 weeks of study entry
* Breast feeding or pregnancy determined by urine pregnancy test in subjects where pregnancy is a possibility (pre-menopausal, sexually active women)
* Subjects with previous allergic reaction to apomorphine or sulfate sensitivity
* Subjects currently taking 5HT3 antagonists

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale of Improvement | Weeks 4 - 8
  Subjects will assess how they feel 30 minutes after taking four doses of drug or placebo.

SECONDARY OUTCOMES:
International RLS Rating Scale (IRLS) | Baseline, 4 weeks, 8 weeks, and 16 weeks
  This is a subjective scale to measure the severity of RLS within the past week.
The Restless Legs Syndrome - 6 Scale (RLS-6) | Baseline, 4 weeks, 8 weeks, and 16 weeks
  This scale measures the severity of daytime versus nighttime RLS symptoms.
Restless Legs Syndrome Quality of Life Questionnaire (RLSQoL) | Baseline, 4 weeks, 8 weeks, and 16 weeks
  This scale assess the quality of life in RLS patients.
Hamilton Depression Scale (HDS) | Baseline, 4 weeks, 8 weeks, and 16 weeks
  This scale assess symptoms of depression.
Epworth Sleepiness Scale (ESS) | Baseline, 4 weeks, 8 weeks, and 16 weeks
  This is a subjective scale that measures a patient's sleepiness.
Clinical Global Impressions - Change | 1 week, 2 weeks, 3 weeks, 4 weeks, 5 weeks, 6 weeks, 8 weeks, 12 weeks, 16 weeks, and 18-20 weeks
  This scale assess how much a patients illness has improved or worsened when compared to a baseline state from the beginning of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: William Ondo, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States